CLINICAL TRIAL: NCT06332430
Title: A Phase 1, Dose Escalation, Open-Label Study of Intratumoral CAN2109 in Subjects With Unresectable or Metastatic Advanced Solid Tumors.
Brief Title: Intratumoral CAN2109 in Subjects With Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Canwell Biotech Limited (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CW-202
Record Dates: First submitted 2024-03-20; First posted 2024-03-27 (Actual); Last update posted 2024-12-19 (Actual); Status verified 2024-12

CONDITIONS: Solid Tumor; Lymphoma
MeSH Terms: conditions — Lymphoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- CAN2109 (Experimental): CAN2109 IT injection every three weeks (Q3W)
  Interventions: Drug: CAN2109

INTERVENTIONS:
Drug: CAN2109 — CAN2109 IT injection (once every 3 weeks)

SUMMARY:
A phase 1, dose escalation, open-label study of intratumoral CAN2109 in subjects with unstable or metastatic advanced solid tumors or lymphomas.

DETAILED DESCRIPTION:
The scope of the study is to evaluate the safety of CAN2109 in humans, explore its safety, efficacy and collect data on the pharmacokinetics, as well as on the pharmacodynamic effect of the drug on the immune system locally and systemically, and on tumor markers.

ELIGIBILITY:
Inclusion Criteria:

1. Able and willing to provide written informed consent and willing to comply with the study's requirements.
2. Male or female age ≥ 18 years at screening.
3. Metastatic or locally advanced solid tumor that has progressed on, is refractory to, or for which there is no efficacious standard of care therapy. Preferred tumor types include the following:

   a. Carcinoma of skin, melanoma, Merkel cell carcinoma (MCC), breast cancer, head and neck squamous cell carcinoma (HNSCC), sarcoma, cervical carcinoma, and colorectal cancer
4. Performance status of 0-1 on the ECOG Performance Scale.

Exclusion Criteria:

1. Unresolved toxicities from prior therapy, defined as having not resolved to Common Terminology Criteria for Adverse Events (CTCAE) Version 5.0 (v5.0) Grade 0 or 1, with exception of endocrinopathies from prior therapy, alopecia, and vitiligo.
2. Treatment with systemic corticosteroids at doses exceeding 10 mg/day prednisone or equivalent.
3. Has an active infection requiring systemic therapy.
4. Unstable/inadequate cardiac function defined as follows:

   1. New York Heart Association Class 3 or 4 congestive heart failure
   2. uncontrolled hypertension
   3. acute coronary syndrome within 6 months
   4. clinical important cardiac arrhythmia
   5. mean corrected QT (QTc) interval corrected for heart rate > 480 ms.
5. A history of interstitial lung disease.
6. A history of coagulopathy resulting in uncontrolled bleeding or other bleeding disorders.
7. Participated in a clinical study of an investigational agent within 30 days of screening.
8. Has known psychiatric, substance abuse, or other disorders that would interfere with cooperation with the requirements of the study in the opinion of the investigator.
9. Is pregnant or breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Estimated)
Dates: Start 2024-05-28 (Actual); Primary Completion 2025-05-30 (Estimated); Study Completion 2026-05-30 (Estimated)

PRIMARY OUTCOMES:
Safety | 12 months
  determined by assessment of dose limiting toxicities per protocol of CAN2109 with cancers.
Recommended Phase 2 Dose (RP2D) | 12 months
  To determine a recommended phase 2 dose of CAN21909 for further development by evaluating number of patients with treatment-related adverse events as assessed by the Common Terminology Criteria for Adverse Events version 5.0 (CTCAE v5.0).
tolerability | 12 months
  determined by assessment of the maximum tolerated dose or maximal assessed dose per protocol of CAN2109 with cancers.

SECONDARY OUTCOMES:
To determine the efficacy of CAN2109 | 12 months
  Proportion of patients experiencing a tumor response or a stable disease according to RECIST 1.1 or iRECIST 1.1 as appropriate.
To evaluate the pharmacodynamics of CAN2109 | 12 months
  Maximum observed plasma and tumor concentration of CAN2109 after IT administration.

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-Sen University Sun Yat-Sen Memorial Hospital, Guangzhou, Guangdong, China